CLINICAL TRIAL: NCT03324555
Title: A Phase 1 Single-ascending Dose Study of the Oral Glucocorticoid Receptor Antagonist ORIC-101 in Healthy Adult Subjects
Brief Title: Study of ORIC-101 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ORIC Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORIC-GR-17001
Record Dates: First submitted 2017-10-25; First posted 2017-10-27 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ORIC-101 (Experimental)
  Interventions: Drug: ORIC-101

INTERVENTIONS:
Drug: ORIC-101 — Oral suspension

SUMMARY:
ORIC-GR-17001 is an open-label, single center, non-randomized, single ascending dose study in healthy male subjects and healthy female subjects of non-child bearing potential. In this study, ORIC-101 will be administered as single-ascending oral doses. The primary objective is to characterize the safety and tolerability of oral ORIC-101.

DETAILED DESCRIPTION:
This is an open-label, single center, non-randomized, single ascending dose study in healthy male subjects and healthy female subjects of non-child bearing potential.

Subjects will receive a single administration of ORIC-101 oral suspension on a single occasion and will be followed in the clinic for at least 96 hours post-dose. Total subject participation will be approximately 5 weeks from screening until discharge from the study.

The primary objective of the study is to characterize the safety and tolerability of oral ORIC-101 administered as a single dose in adult healthy subjects. The secondary objective of the study is to evaluate the pharmacokinetics of ORIC-101 and its metabolites M1 and M2. The exploratory objective of the study is to assess the pharmacodynamics of ORIC-101 by measurement of serum and urine levels of cortisol and other biological markers in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or healthy females of non-child bearing potential
2. Age 18 to 55 years, inclusive
3. Weighs more than 50 kilograms (kg), and less than 120 kg, with a body mass index of 18.0 to 32.0 kg/meters squared

Exclusion Criteria:

1. Subjects who have received any investigational medicinal product (IMP) in a clinical research study within 5 half-lives or within 45 days prior to first dose. However, in no event, shall the time between last receipt of IMP and first dose be less than 30 days
2. History of any drug or alcohol abuse in the past 2 years
3. Current smokers and those who have smoked within the last 12 months
4. Females of childbearing potential (female subjects must have a negative pregnancy test). A woman is considered of childbearing potential unless she is permanently sterile (hysterectomy, bilateral salpingectomy, tubal ligation or bilateral oophorectomy) or is postmenopausal (had no menses for 12 months without an alternative medical cause and a serum follicle-stimulating hormone [FSH] concentration ≥40 international units per litre (IU/L))
5. Women with a history of unexplained vaginal bleeding or endometrial hyperplasia with atypia or endometrial carcinoma
6. Current disease requiring treatment with systemic corticosteroids.
7. Serious adverse reaction or serious hypersensitivity to mifepristone, or any other drug, or the formulation excipients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability, as assessed by incidence and severity of adverse events. | 96 hours post-dose

SECONDARY OUTCOMES:
Pharmacokinetics, as assessed by time of observed maximum concentration (Tmax) | 96 hours post-dose
Pharmacokinetics, as assessed by maximum concentration observed (Cmax) | 96 hours post-dose
Pharmacokinetics, as assessed by area under the concentration versus time curve from time 0 to 24 hours post-dose (AUC(0-24)) | 96 hours post-dose
Pharmacokinetics, as assessed by area under the concentration versus time curve from time 0 to last measurable concentration (AUC(0-last)) | 96 hours post-dose
Pharmacokinetics, as assessed by area under the concentration versus time curve from time 0 extrapolated to infinity (AUC(0-inf)) | 96 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Research Center, Miami, Florida, United States